CLINICAL TRIAL: NCT02838277
Title: Insight Into Subcutaneous Adipose Tissue Disorders As Part of The TREAT Program (Treatment, Research, Education, Adipose Tissue) at the University of Arizona
Brief Title: Insight Into Subcutaneous Adipose Tissue Disorders
Acronym: INSIGHT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: Lipedema Foundation (Other)
Responsible Party: Principal Investigator, KHerbst, Associate Professor, University of Arizona
Other Study IDs: 1602399502A001
Record Dates: First submitted 2016-06-28; First posted 2016-07-20 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Lipedema; Dercum's Disease; Familial Multiple Lipomatosis; Madelung's Disease
Keywords: lymphatic vessels; leaky vessels; hypertrophic adipocyte
MeSH Terms: conditions — Lipedema; Adiposis Dolorosa; Familial Multiple Lipomatosis; Lipomatosis, Multiple Symmetrical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, adipose tissue and DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Lipedema: Women with all stages of lipedema
- Dercum's disease: Men and women with nodular, mixed and diffuse Dercum's disease
- Control: Sex, age and BMI matched controls.
- Familial Multiple Lipomatosis: Women and men with multiple lipomas and/or angiolipomas
- Madelung's disease: Men and women with different types of Madelung's disease.

SUMMARY:
The INSIGHT study aims to phenotype individuals with subcutaneous adipose tissue (SAT) disorders specifically lipedema and Dercum's disease with an aim to find a cure for the SAT in these disorders that is resistant to diet and exercise.

DETAILED DESCRIPTION:
Lipedema is a syndrome of painful fatty enlargement of the buttocks, hips and thighs primarily in women which cannot be lost by diet, exercise or bariatric surgery. Arms are affected in 80% of women with lipedema to varying degrees. The etiology of lipedema is not known and there are no evidence-based treatments that work for a majority of individuals except for excision of the subcutaneous adipose tissue (SAT) by liposuction which has risks. Millions of women are affected with lipedema yet they are grossly under-diagnosed, have mobility issues and can develop lymphedema. The goal of this project is to better understand the etiology of lipedema SAT, find out how it is different from non-lipedema SAT, to improve our ability to identify the abnormal SAT and determine the response of the tissue to therapeutics by imaging and biomarkers. People with diffuse Dercum's disease (DD) appear to have lipedema plus a tissue inflammation that causes illness and pain. People with SAT disorders that have similarities to lipedema will also be included in this protocol. More research is needed to determine how these fatty disorders are similar and different from each other and from obesity so they can be distinguished clinically and by laboratory testing and imaging. Since these painful fatty disorders are associated with SAT growth, research focused on these disorders may provide unique insight into mechanisms of obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory males and/or females of any race able to understand the consent process.
2. 19-70 years of age.
3. Diagnosis of lipedema, Dercum's disease or familial multiple lipomatosis or other similar fat disorder.
4. Individuals without a fat disorder (will be matched by age, sex, race and body mass index to individuals in "2").
5. Weight stable for past three months within a 10 pound range per personal report of the subject.
6. Overweight or obese (BMI > 26 kg/m2) in order to be able to get enough SAT for the biopsy.
7. Individuals with BMI < 26 kg/m2 may participate in all aspects of the study protocol except the SAT biopsy.
8. Thyroid levels in the normal range as confirmed by a TSH level. May have treated hypothyroidism that is stable over 6 months.

Exclusion Criteria:

1. HIV infection (because of the associated lipodystrophy and fatty growths [lipomas]).
2. Subjects will be excluded from having a SAT biopsy with any history of scleroderma, keloid formation or other skin condition that would result in substantial scarring after biopsy, a history of recurrent cellulitis, any history of bleeding diathesis that would place the subject at great risk for persistent bleeding after a biopsy/liposuction, any history of major complication after a previous biopsy including requirement of a blood transfusion, hospitalization, failure to heal, or major infection, requiring intravenous antibiotics, or anyone whose skin and tissue would put them at risk for an infection after the biopsy per the assessment of study staff and the principal investigator. These individuals may participate in the remainder of the protocol, just not the SAT biopsy.
3. Use of any immunosuppressant or corticosteroid medication.
4. Use of any anti-inflammatory medication such as NSAIDs, aspirin, histamine (H) 1 blocker, H2 blocker, tetracycline or corticosteroids within five days of the study procedure visit.
5. Use of medications that might cause weight gain (e.g., second generation anti-psychotics).
6. Blood donation less than 56 days prior to screening visit.
7. Tobacco or marijuana use which may alter inflammation in the body.
8. Any antibiotics within the last month.
9. Barium enema in the last week which would affect gut bacteria and the MRI.
10. Pregnancy due to the risks associated with the fat biopsy in the area of the fetus and because pregnancy will alter hormone levels.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women with lipedema and Dercum's disease and controls.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Transcriptomics of all enrolled subjects from a single timepoint to assess for changes in gene expression in lipedema tissue compared to controls | Single time point study with imaging, blood draw, exam and biopsies over multiple days for a total of approximately 8 hours time.
  This is a phenotyping study that collects data as a single time point though studies may occur on different days.
Metabolomics of all enrolled subjects from a single timepoint to assess for changes in metabolites in lipedema tissue compared to controls | Single time point study with imaging, blood draw, exam and biopsies over multiple days for a total of approximately 8 hours time.
  This is a phenotyping study that collects data as a single time point though studies may occur on different days.
Lipidomics of all enrolled subjects from a single timepoint to assess for changes in lipid particles in lipedema tissue and blood compared to controls | Single time point study with imaging, blood draw, exam and biopsies over multiple days for a total of approximately 8 hours time.
  This is a phenotyping study that collects data as a single time point though studies may occur on different days.
Cytokines of all enrolled subjects from a single timepoint to assess for changes in cytokine arrays in lipedema tissue and blood compared to controls | Single time point study with imaging, blood draw, exam and biopsies over multiple days for a total of approximately 8 hours time.
  This is a phenotyping study that collects data as a single time point though studies may occur on different days.
Myostatin of all enrolled subjects from a single timepoint to assess for levels of myostatin in lipedema tissue and blood compared to controls | Single time point study with imaging, blood draw, exam and biopsies over multiple days for a total of approximately 8 hours time.
  This is a phenotyping study that collects data as a single time point though studies may occur on different days.

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Herbst, PhD, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona College of Medicine (South Campus), Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared with investigators who submit a request.

REFERENCES:
- [Derived] Allen M, Schwartz M, Herbst KL. Interstitial Fluid in Lipedema and Control Skin. Womens Health Rep (New Rochelle). 2020 Oct 14;1(1):480-487. doi: 10.1089/whr.2020.0086. eCollection 2020. PMID 33786515